CLINICAL TRIAL: NCT03825458
Title: Creation of a Cohort for the Quantitation and Characterization of Circulating Viral RNAs as a New Biomarker of Hepatitis B Functional Cure.
Acronym: CirB-RNA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0436; 2018-A02558-47 (Other: ID-RCB)
Record Dates: First submitted 2018-12-31; First posted 2019-01-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma EDTA and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling — Blood sampling at each clinical follow-up visit.

SUMMARY:
The " CirB-RNA " cohort aims to create a biological collection associated with clinical and biological data from patients with hepatitis B infection. This project is part of a much larger program that aims to characterize and quantify circulating viral RNAs as a possible new biomarker of hepatitis B functional cure.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients and minor children over 6 years of age (in Lyon) with acute or chronic hepatitis B or presenting with HBsAg loss (with/without HBs seroconversion). (Co-infected patients with HDV and/or HCV and/or HIV are eligible)
* Patients requiring blood sampling for medical care at the time of the medical appointment.
* Informed patients who do not refuse to participate.
* Persons not affiliated to a social security scheme and persons receiving medical assistance from the state may be asked to participate in the study

Exclusion Criteria:

* Patients participating at the time of the inclusion to an interventional trial evaluating a drug likely to interfere with this study.
* Persons deprived of their liberty by a judicial or administrative decision
* Adults who are subject to a legal protection measure
* Children less than 6 years old (in Lyon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatitis B infection (acute or chronic) or presenting with HBsAg loss (with/without anti-HBs seroconversion).
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2029-06-25 (Estimated); Study Completion 2029-06-25 (Estimated)

PRIMARY OUTCOMES:
Number of plot samples collected | maximum 46 months
  The aim of this study is the constitution of a cohort with biological collection associated with clinical and biological data Data and samples will be collected at each follow-up visit until end of project (longitudinal study).
  This cohort is the first step of a research program and will be use in further study which are part of this research program. All studies of this research program aim to improve knowledge about hepatitis B, develop and validate a new biomarker of hepatitis B cure.

CONTACTS AND LOCATIONS:
Locations (6):
- France (3):
  - Hepatology department - Groupement Hospitalier Nord - Hôpital de la Croix-Rousse, Lyon
  - Hôpital de la Croix-Rousse - Service de maladies infectieuses et tropicales, Lyon
  - Department of Hepato-gastroenterology and pediatric nutrition - Hôpital Femme-Mère Enfant, Lyon
- Italy (3):
  - Gastroenterology and Hepatology department - • Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Gastroenterology and Hepatology department - • Università degli Studi di Palermo, Palermo
  - Infectious diseases and hepatology unit - Azienda Ospedaliero, Parma

IPD SHARING:
Plan to Share IPD: No